CLINICAL TRIAL: NCT01796782
Title: A Prospective, Randomized, Open-label, Phase II Study of QYHJ Granules Versus Xeloda in the Second-line Treatment of Patients With Metastatic Pancreatic Cancer
Brief Title: QYHJ Granules Versus Xeloda in Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, liu lu ming, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCM-002
Record Dates: First submitted 2012-12-16; First posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xeloda (Active Comparator): Subjects will receive Xeloda until progression
  Interventions: Drug: Xeloda
- QYHJ Granules (Experimental): patients will receive QYHJ Granules until progression
  Interventions: Drug: QYHJ Granules

INTERVENTIONS:
Drug: Xeloda — Xeloda dose is calculated according to body surface area.The recommended dose is 1000 mg/m² administered orally twice daily (morning and evening; equivalent to 2000 mg/m² total daily dose) for 2 weeks followed by a 1-week rest period given as 3-week cycles
  Other Names: Capecitabine
  Arms: Xeloda
Drug: QYHJ Granules — 1-4 bags bid , days 1-42, every 6 weeks
  Arms: QYHJ Granules

SUMMARY:
Primary End Point:

- To compare the overall survival (OS) using QYHJ Granules or Xeloda as the second therapy in patients with metastatic pancreatic cancer.

Secondary End Points:

* Compare clinical efficacy by other measures including PFS,tumor response,and changes in quality of life (QOL) between these two groups.
* Examine the feasibility and assess the side effects of treatment using QYHJ Granules in patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed metastatic pancreatic adenocarcinoma.
* Patients have failed from the prior chemotherapy without Xeloda. Adjuvant chemotherapy containing Xeloda and 6 months before recruitment is included.
* Patients haven't taken QYHJ Granules before. Prior exposure to Traditional Chinese Medicine not based on QYHJ Formula is allowed provided that at least one week washout time is given prior to initiation of experimental treatment.
* ECOG performance status 0, 1 or 2.
* Measurable disease by RECIST criteria must be present. Bone scan abnormalities alone will not be accepted as measurable disease. Lytic lesions seen on plain radiographs will not be accepted as measurable disease but will be evaluated in conjunction with bone scan abnormalities. Pure blastic bone metastases will not be accepted as measurable disease. Pleural or peritoneal effusions will not be accepted as measurable disease. Irradiated lesions are not considered measurable.
* Patients must not be pregnant. Serum beta-HCG will be checked in all premenopausal patients.
* Patients must have adequate organ functions reflected by the laboratory criteria below: neutrophil counts ≥ 1.5×109 /L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 85 g/L, Serum creatinine < 2.0 mg/dL, Bilirubin < 1.5 mg/dL, ALT < 3 x normal, albumin >30g/L.
* Age ≥ 18.
* Prior local therapy, e.g., TACE or radiation, is allowed provided that at least 4 weeks washout time is given.
* Concomitant bisphosphonates are allowed for patients with bone metastases. Patients with jaundice must have a biliary drainage decompression operation before recruitment.
* Ability to understand and the willingness to sign a written informed consent.
* Subjects who have a life expectancy of at least 3 months.

Exclusion Criteria:

* ECOG performance status 3 or 4.
* Known central nervous system involvement and leptomeningeal disease.
* Previous Xeloda-based chemotherapy （except usage for Adjuvant chemotherapy and 6 months before recruitment）.
* Prior treatment with QYHJ Granules.
* Other serious illness or condition including cardiac disease including congestive heart failure (New York Heart Association Classification III or IV),unstable angina, myocardial infarction within the past six months, severe arrhythmia.
* Concurrent infection requiring intravenous antibiotics, active HIV infection/HIV disease, psychiatric disorders, drug abuse.
* Known allergies to the QYHJ or Xeloda.
* Pregnant or lactating females. Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days with a confirmatory urine pregnancy test within 7 days prior to study treatment start. Men and women of childbearing potential not using effective means of contraception.
* Known other non-adenocarcinoma pathological type.
* Other primary tumour (including primary brain tumours) within the last 5 years prior to enrollment, except for adequately treated carcinoma in situ of the cervix or basal cell skin cancer.
* Inability to take oral medication, prior surgical procedures affecting absorption or unwilling to take the Traditional Chinese Medicine.
* Patiens who are suffering from diarrhea.
* Subjects with poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | up to 3 years

SECONDARY OUTCOMES:
Progression free survival（PFS） | up to 3 years
Tumor response（ORR、DCR） | up to 3 years
Clinical benefit rate （CBR）and QOL assessment | up to 3 years
Number of adverse events of QYHJ Formula | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: zhen Chen, M.D., Principal Investigator — Fudan University; lu ming Liu, M.D., Study Director — Fudan University